CLINICAL TRIAL: NCT04765527
Title: Nutritional-Based Strategy to Counter Exercise-Induced Muscle Damage and OxInflammation
Brief Title: Turmeric and Exercise-Induced Muscle Damage and Oxinflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: MegaFood (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-0294
Record Dates: First submitted 2020-10-16; First posted 2021-02-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Muscular Injury
Keywords: turmeric; muscular strength; inflammation; exercise; oxidative stress
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group
Who Masked: Participant, Investigator
Masking Description: Coded, capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turmeric (Experimental): Dietary supplement, Turmeric Strength for Joint, containing turmeric root extract (with 350 mg curcumin), black pepper extract, boswellia gum resin extract, devil's claw root extract, and ginger root; 2 tablets each day in the morning prior to breakfast, 2 weeks, and Monday through Friday of exercise and recovery.
  Interventions: Dietary Supplement: Turmeric Strength for Joint
- Placebo (Placebo Comparator): Placebo tablets; 2 tablets each day in the morning prior to breakfast, 2 weeks, and Monday through Friday of exercise and recovery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Turmeric Strength for Joint — Turmeric-based tablets
  Other Names: Turmeric
  Arms: Turmeric
Dietary Supplement: Placebo — Placebo tablets
  Other Names: Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the effect of using a turmeric-based supplement for 2-weeks on muscle damage and soreness that occur in the body after 90-minutes of exercise. Participants will first come to the human performance lab (HPL) for orientation and pre-study fitness tests including muscular fitness and body composition. Participants will be randomized to turmeric or placebo groups, and take 2 tablets of the supplements each day for the first two weeks. Participants will report back to the HPL on a Monday to engage in weight lifting and calisthenics for 90 minutes. Fitness tests (vertical jump, bench press, leg-back lift for strength, 30-second cycling sprint test) and blood samples will be given and collected before and after this exercise session. Participants will then come back to the HPL each morning, Tuesday through Friday, in the early morning to provide blood samples and retake the fitness tests. This study will entail seven HPL visits over a 3-week period.

DETAILED DESCRIPTION:
Orientation, Supplementation, and Basic Study Procedures (Visit #1): Participants will first come to the Human Performance Lab (600 Laureate Way, North Carolina Research Campus, Kannapolis, NC) for an orientation to study procedures. This will include a review of the consent form, completion of basic questionnaires, and an introduction to the eccentric muscle exercise bout and the strength/power performance testing protocol (about 1.5 hours) (visit #1). This will be followed by another lab session for pre-study measurements and sample collection (visit #2). Participants will be randomized to turmeric or placebo groups, and provided a 2-weeks supply of supplements (in supplement trays). Participants will consume 2 tablets each day in the morning just prior to breakfast. The supplement and placebo tablets will look the same. The supplements will have codes. Participants and the staff will not know what are in the tablets until the study is over. The supplement is called "Turmeric Strength for Joint" and is sold by the study sponsor (MegaFood). For purposes of this study, the supplement will be called "turmeric". The ingredients are healthy and include turmeric root extract, black pepper extract, boswellia gum resin extract, devil's claw root extract, and ginger root. The turmeric supplement provides a minimum of 300 mg curcumin. Compliance to the supplement plan will be checked weekly through email correspondence from the Research Manager. A 3-day food record will be collected during the end of the 2-week supplementation period to assess the participants' background diet.

The study will include 5 other lab visits during a one-week period starting on a Monday (visit #3), with morning visits at about 7:00 am on Tuesday through Friday (visits 4-7). At each of the 7 lab visits, participants will come to the lab at 7:00 am not having consumed food or beverages (other than water) for at least the previous 9 hours, and having abstained from vigorous exercise for at least the previous 24-48 hours. The Monday session will take about 2.5 hours (7:00 to 9:30 am), and the Tuesday through Friday sessions will take about 30-45 minutes each. The total amount of time participants will be asked to volunteer for this study is about 8-9 hours at the performance lab. Seven blood samples will be collected and analyzed for various measures of muscle damage, inflammation, and oxidative stress. After each of the blood draws, participants will complete the Profile of Mood States (POMS) questionnaire to gauge mood, energy, and vitality. Participants will also provide a delayed onset of muscle soreness (DOMS) rating. Two urine samples will be collected (before and after the 2-week supplementary period) and analyzed for key metabolic markers of turmeric ingestion.

Baseline Testing (Visit #2) Participants will come to the lab at 7:00 am in an overnight fasted state dressed in exercise clothes. Participants will provide a blood sample. A trained phlebotomist will collect a maximum of 35 ml blood (a little over 2 tablespoons). Participants will also provide a spot urine sample in a private location in the restroom. Participants will collect a mid-stream urine sample in a disposable urine cup. Height, body weight, and body composition will be measured in a private section of the lab. Bioelectrical impedance (BIA) using the seca BIA scale will be used to assess body composition (i.e., the percent of body weight that is fat tissue) and body weight. Participants will remove shoes and socks and stand with bare feet on the seca scale for about 7-10 seconds while grasping side rails with their hands. Percent body fat will also be measured using the BodPod. Participants will sit inside the BodPod with a tight-fitting swim suit for about 10 minutes while body fat is calculated.

The Profile of Mood States (POMS) (short version, 40 items) is a rating scale to assess "right now" mood states, energy, and vitality. Participants will also provide a rating of delayed onset of muscle soreness (DOMS) using a 1-10 scale.

Participants will perform some light exercises to warm up, followed by four muscle function tests: vertical jump, bench press, leg-back strength, and anaerobic power through the 30-second Wingate test.

1. Vertical jump: Participants will first stand erect with the feet flat on the floor and reach as high as possible with both arms and hands (standing reach height). Participants will then squat down and jump as high as possible with one arm and hand, and tap the measuring device on the Vertec vertical jump apparatus (jump height). This will be repeated three times, with the best score recorded as the difference between the jump and standing reach heights.
2. Bench press to exhaustion: Participants will lie down supine on a bench, and with spotters standing on either side attempt to bench press a weighted bar equal to 50% (females) or 75% (males) body weight as many times as possible (to a metronome set at 60 beats/min or 30 lifts/min). The bar must touch a foam block on the chest lightly in the down position, and the arms must be straight in the up position.
3. Leg-Back Strength: Leg/lower back strength will be assessed with a dynamometer. With the legs slightly bent at the knee, participants will grasp a bar attached via a chain and a force measuring device with straight arms, and then lift up with maximal effort for several seconds. This will measure the isometric strength of both legs and back, and will be repeated three times.
4. 30-Second Wingate Cycling Test: The Lode cycle ergometer will be adjusted to body weight (7 watts per kilogram), and then participants will sprint cycle at maximal speed for 30 seconds. The peak power and average power will be recorded and adjusted to body mass.

Testing Sequence, Day of Eccentric Muscle Exercise (Monday, Visit #3) and 4-Days Recovery (Tuesday through Friday) (Visits #4-7):

Participants will come to the lab at 7:00 am in an overnight fasted state (i.e., no food or beverages other than water for at least the previous 9 hours). Participants will be weighed and then provide a blood sample. A spot urine sample will be collected on Monday. Participants will then complete the POMS questionnaire, and give a DOMS rating. The supplements will be consumed with water. Participants will perform some light exercises to warm up, followed by the four muscle function tests: vertical jump, bench press, leg-back strength, and anaerobic power through the 30-second Wingate test. Participants will take these performance tests before and after the 90-minute eccentric muscle exercise bout, and each of the following four mornings at the performance lab.

After taking the four performance tests, participants will engage in 90-minutes of eccentric exercise that include 16 movements (calisthenics, resistance exercise, jumps, 2-3 sets, with rest intervals).

Immediately following exercise, participants will provide a blood sample, complete the POMS questionnaire, and provide a DOMS muscle soreness rating. Participants will then take the four muscle function tests. Participants will return at 7:00 am in an overnight fasted state four days in a row (Tuesday through Friday) after Monday's eccentric exercise bout, and provide a blood sample, complete the POMS, provide DOMS ratings, and follow this with ingestion of the supplements. Following ingestion of the supplements, participants will take the four muscle function tests. During this week of testing and recovery, participants will engage in normal training and diet habits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18-50 years.
* Non-smoker.
* Body mass index less than 35 kg/m2 (below moderate or severe obesity).
* Not engaged in regular resistance training (less than 3 sessions per week).
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, protein supplements, herbs, and medications that influence inflammation and immune function (especially Advil, Motrin, aspirin, and similar anti-inflammatory drugs) for the duration of the study. (You will review your supplement and medication use with the Research Manager during orientation).
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.

Exclusion Criteria:

* Inability to comply with study requirements.
* Engaged in regular resistance training (3 or more sessions per week, on average).
* Body weight below 110 pounds.
* Pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* History of allergic reactions to turmeric, devil's claw, boswellia extract, or ginger extract.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Serum concentration of creatine kinase | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle damage biomarker

SECONDARY OUTCOMES:
Serum concentration of myoglobin | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle damage markers
Rating of Delayed onset of muscle soreness | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Self-reported perception of muscle soreness, 1-10 scale, with 1=no soreness to 10=extremely sore
Plasma concentration of 4-hydroxynonenal (4HNE) | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Oxidative stress biomarkers
Serum concentration of C-reactive protein | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Inflammation biomarker
Plasma concentration of IL-6 | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Inflammation biomarkers
Serum concentration of cortisol | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Stress hormone
Urine concentration of curcuminoid metabolites | Change from pre-to-post-supplementation, 2 week period
  Curcumin metabolites: tetrahydrocurcumin (THC), hexahydrocurcumin (HHC), and octahydrocurcumin (OHC)
Vertical jump height | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Vertical jump height as a muscle function test
Bench press repetitions | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle performance, bench press to exhaustion with weighted bar
Leg-back strength kilograms | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle performance, leg-back strength with a dynamometer
30-second Wingate cycle test watts | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Anaerobic sprint power cycling test, peak and average watts
Rating of Profile of Mood States (POMS) | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Rating scale to assess mood states, energy, vitality; 0 to 4 scale, with 0=not at all to 4=extremely

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Will provide basic data spreadsheet upon request.